CLINICAL TRIAL: NCT04217551
Title: Influence of Cooling Duration on Efficacy in Cardiac Arrest Patients - A Multicenter, Randomized, Adaptive Clinical Trial to Identify the Optimal Duration of Induced Hypothermia for Neuroprotection in Comatose Survivors of Cardiac Arrest
Brief Title: Influence of Cooling Duration on Efficacy in Cardiac Arrest Patients
Acronym: ICECAP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Johns Hopkins University (Other); Medical University of South Carolina (Other); National Institutes of Health (NIH) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, William J Meurer, Associate Professor of Emergency Medicine and Neurology, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: G160072; U01NS073476 (NIH)
Record Dates: First submitted 2019-12-30; First posted 2020-01-03 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Cardiac Arrest, Out-Of-Hospital; Hypothermia, Induced; Hypoxia-Ischemia, Brain
Keywords: Bayesian Adaptive Clinical Trial; Hypothermia, therapeutic; Coma
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Hypothermia; Hypoxia-Ischemia, Brain; Coma | interventions — Hypothermia, Induced

STUDY DESIGN:
Intervention Model Description: Bayesian Adaptive Design
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessors will be blinded to the treatment assignment of the participant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (20):
- 6 hours - shockable (Experimental): Participants with shockable initial rhythm will be assigned to receive 6 hours of hypothermia with a target of 33 degrees followed by 6 hours of controlled rewarming.
  Interventions: Device: Therapeutic Hypothermia
- 12 hours - shockable (Experimental): Participants with shockable initial rhythm will be assigned to receive 12 hours of hypothermia with a target of 33 degrees followed by 12 hours of controlled rewarming.
  Interventions: Device: Therapeutic Hypothermia
- 18 hours - shockable (Experimental): Participants with shockable initial rhythm will be assigned to receive 18 hours of hypothermia with a target of 33 degrees followed by 18 hours of controlled rewarming.
  Interventions: Device: Therapeutic Hypothermia
- 24 hours - shockable (Experimental): Participants with shockable initial rhythm will be assigned to receive 24 hours of hypothermia with a target of 33 degrees followed by 24 hours of controlled rewarming.
  Interventions: Device: Therapeutic Hypothermia
- 30 hours - shockable (Experimental): Participants with shockable initial rhythm will be assigned to receive 30 hours of hypothermia with a target of 33 degrees followed by 24 hours of controlled rewarming.
  Interventions: Device: Therapeutic Hypothermia
- 36 hours - shockable (Experimental): Participants with shockable initial rhythm will be assigned to receive 36 hours of hypothermia with a target of 33 degrees followed by 24 hours of controlled rewarming.
  Interventions: Device: Therapeutic Hypothermia
- 42 Hours - shockable (Experimental): Participants with shockable initial rhythm will be assigned to receive 42 hours of hypothermia with a target of 33 degrees followed by 24 hours of controlled rewarming.
  Interventions: Device: Therapeutic Hypothermia
- 48 hours - shockable (Experimental): Participants with shockable initial rhythm will be assigned to receive 48 hours of hypothermia with a target of 33 degrees followed by 24 hours of controlled rewarming.
  Interventions: Device: Therapeutic Hypothermia
- 60 hours - shockable (Experimental): Participants with shockable initial rhythm will be assigned to receive 60 hours of hypothermia with a target of 33 degrees followed by 24 hours of controlled rewarming.
  Interventions: Device: Therapeutic Hypothermia
- 72 hours - shockable (Experimental): Participants with shockable initial rhythm will be assigned to receive 72 hours of hypothermia with a target of 33 degrees followed by 24 hours of controlled rewarming.
  Interventions: Device: Therapeutic Hypothermia
- 6 hours - non shockable (Experimental): Participants with non-shockable initial rhythm will be assigned to receive 6 hours of hypothermia with a target of 33 degrees followed by 6 hours of controlled rewarming.
  Interventions: Device: Therapeutic Hypothermia
- 12 hours - non-shockable (Experimental): Participants with non-shockable initial rhythm will be assigned to receive 12 hours of hypothermia with a target of 33 degrees followed by 12 hours of controlled rewarming.
  Interventions: Device: Therapeutic Hypothermia
- 18 hours - non-shockable (Experimental): Participants with non-shockable initial rhythm will be assigned to receive 18 hours of hypothermia with a target of 33 degrees followed by 18 hours of controlled rewarming.
  Interventions: Device: Therapeutic Hypothermia
- 24 hour - non-shockable (Experimental): Participants with non-shockable initial rhythm will be assigned to receive 24 hours of hypothermia with a target of 33 degrees followed by 24 hours of controlled rewarming.
  Interventions: Device: Therapeutic Hypothermia
- 30 hours - non-shockable (Experimental): Participants with non-shockable initial rhythm will be assigned to receive 30 hours of hypothermia with a target of 33 degrees followed by 24 hours of controlled rewarming.
  Interventions: Device: Therapeutic Hypothermia
- 36 hours - non-shockable (Experimental): Participants with non-shockable initial rhythm will be assigned to receive 36 hours of hypothermia with a target of 33 degrees followed by 24 hours of controlled rewarming.
  Interventions: Device: Therapeutic Hypothermia
- 42 hours - non-shockable (Experimental): Participants with non-shockable initial rhythm will be assigned to receive 42 hours of hypothermia with a target of 33 degrees followed by 24 hours of controlled rewarming.
  Interventions: Device: Therapeutic Hypothermia
- 48 hours - non-shockable (Experimental): Participants with non-shockable initial rhythm will be assigned to receive 48 hours of hypothermia with a target of 33 degrees followed by 24 hours of controlled rewarming.
  Interventions: Device: Therapeutic Hypothermia
- 60 hours - non-shockable (Experimental): Participants with non-shockable initial rhythm will be assigned to receive 60 hours of hypothermia with a target of 33 degrees followed by 24 hours of controlled rewarming.
  Interventions: Device: Therapeutic Hypothermia
- 72 hours - non-shockable (Experimental): Participants with non-shockable initial rhythm will be assigned to receive 72 hours of hypothermia with a target of 33 degrees followed by 24 hours of controlled rewarming.
  Interventions: Device: Therapeutic Hypothermia

INTERVENTIONS:
Device: Therapeutic Hypothermia — Participants will receive therapeutic hypothermia for the assigned number of hours with controlled rewarming, using a closed-loop temperature control device.

SUMMARY:
A multicenter, randomized, adaptive allocation clinical trial to determine if increasing durations of induced hypothermia are associated with an increasing rate of good neurological outcomes and to identify the optimal duration of induced hypothermia for neuroprotection in comatose survivors of cardiac arrest.

DETAILED DESCRIPTION:
A multicenter, randomized, adaptive allocation clinical trial to determine if increasing durations of induced hypothermia are associated with an increasing rate of good neurological outcomes and to identify the optimal duration of induced hypothermia for neuroprotection in comatose survivors of cardiac arrest.

Cardiac arrest is a common and devastating emergency of the heart and the brain. More than 380,000 patients suffer out of hospital cardiac arrest (OHCA) each year in the US. Improvements in cardiac resuscitation (the early links in the "chain of survival" for patients with OHCA) are tempered by our limited ability to resuscitate and protect the brain from global cerebral ischemia.

Neurological death and disability are common outcomes in survivors of cardiac arrest. Therapeutic cooling of comatose patients resuscitated from shockable rhythms markedly increases the rate of good neurological outcome, but poor outcomes still occur in as many as 50%, and the benefit of cooling in those resuscitated from asystole and pulseless electrical activity has not been shown in a randomized study.

Objectives:

The overarching goal of this project is to identify clinical strategies that will increase the number of patients with good neurological recovery from cardiac arrest. We hypothesize that longer durations of cooling may improve either the proportion of patients that attain a good neurological recovery or may result in better recovery among the proportion already categorized as having good outcomes.

Primary Objectives:

A. To determine, in each of two populations of adult comatose survivors of cardiac arrest (those with initial shockable rhythms and those with pulseless electrical activity (PEA)/asystole), the shortest duration of cooling that provides the maximum treatment effect as determined by a weighted 90 day modified Rankin score B. To determine, in each of two populations of adult comatose survivors of cardiac arrest (those with initial shockable rhythms and those with PEA/asystole), whether increasing durations of cooling are associated with better outcomes or recovery implying efficacy of hypothermia to no cooling.

Secondary Objectives:

To characterize the overall safety and adverse events associated with duration of cooling To characterize the effect of duration of cooling on neuropsychological outcomes To characterize the effect of duration of cooling on patient reported quality of life

Design:

This study is a randomized, response-adaptive, duration (dose) finding, comparative effectiveness clinical trial with blinded outcome assessment. The design is based on a statistical model of response as defined by the primary endpoint, a weighted 90-day mRS, across the treatment arms. The design will fit patient outcome data to a duration response model (separately for shockable and non-shockable rhythms), in which the potentially non-linear association between durations of cooling and the primary endpoint are estimated. All conclusions about the treatment arms are based on this model. The functional form of the duration-response model is flexible and able to fit many different shapes for the duration-response curve. Specifically it is parameterized to identify up to two change-points in the treatment effect across arms, allowing it to fit an increasing, decreasing, flat, plateau, or U-shape duration-response curve.

Subjects will initially be equally randomized between 12, 24, and 48 hours of cooling. After the first 200 subjects have been randomized, additional treatment arms between 12 and 48 hours will be opened and patients will be allocated, within each rhythm type, by response adaptive randomization. As the trial continues, shorter and longer duration arms may be opened. Specifically, a 6-hour duration arm will be opened if the emerging duration-response curve from 12 hours is flat. Similarly, a 60-hour or 72-hour duration arm will be opened if the emerging duration response curve shows an increasing treatment benefit through 48 hours.

This trial will have frequent interim analyses to stop the trial early for futility if it is highly likely that no treatment arm offers a greater benefit then the 6-hour duration arm.

Primary Outcome Measure:

The primary outcome measure will be the modified Rankin scale at 90 days after return of spontaneous circulation. The mRS will be analyzed as a weighted score incorporating both the proportion of subjects achieving a good neurological outcome and degree of residual functional impairment among those with good neurological outcomes.

Study Population:

Comatose adult survivors of out of hospital cardiac arrest that have already been rapidly cooled using a definitive temperature control method (endovascular or surface) will be enrolled in the emergency department or intensive care unit. Hub and spoke hospitals from the SIREN network will be enriched with high potential ancillary Hubs. Approximately 50 hospitals are anticipated to each enroll an average of 9 subjects per year.

Randomization:

Central computerized randomization by web-based interface will be used. Subjects will be potentially randomized over the course of the trial to the following possible durations of cooling (in hours): 6, 12, 18, 24, 30, 36, 42, 48, 60, and 72. The first 200 patients will be randomized 1:1:1 to the 12, 24, and 48-hour durations only. After this initial "burn in" period, response adaptive randomization will be used to allocate subjects to durations inclusive of 12 to 48 hours initially, and then subsequently to the 6, 60 or 72 hour durations if specified conditions are met and the emerging duration-response curve suggests that the maximum treatment benefit might be on those durations. The response adaptive randomization probabilities for each arm will be determined separately for the two rhythm type populations. Randomization probabilities will be updated monthly, or approximately every 38 patients based on the expected accrual rate.

Consent:

Eligible patients for this trial will not have capacity to provide informed consent. Written informed consent from a legally authorized representative will be required.

Intervention:

The intervention will be random allocation to duration of cooling after cardiac arrest. Cooling in the study will be by a definitive temperature control method to a target temperature of 33 deg C. Any endovascular or surface cooling system with closed loop feedback will be allowed. Duration of cooling will be measured from the time that cooling with a definitive device is initiated in the hospital. As part of routine medical care, cooling may be initiated by emergency medical service (EMS) or in the emergency department. Eligibility will require that a temperature of <34 degrees C be obtained by 240 minutes after cardiac arrest. After the allocated duration of cooling is completed, controlled rewarming will be performed. Rewarming to a temperature of 36.5 deg C will occur over the shorter of 24 hours or a rewarming period equal to the allocated duration of cooling. Definitive cooling devices may be used for maintenance of normothermia after rewarming is complete. A clinical standardization guideline will be followed to reduce the effects of practice variability. Key physiologic and practice variables will be tracked and compliance with clinical standardization and deviation from physiologic targets reported back to study teams.

Statistical Analysis for the Primary Outcome Measure:

We will model the mean weighted mRS at 90 days across the treatment arms. The weighted mRS incorporates both the proportion of subjects achieving a good neurological outcome and degree of impairment among those with good neurological outcomes. The primary analysis is conducted separately for each rhythm type, allowing for a different treatment effect by rhythm type, and has two components. First, we identify the most likely target duration, where the target duration is the shortest duration that achieves the maximum treatment effect (Objective A). Second, we calculate whether the efficacy of any duration is superior to any shorter duration of cooling indicating a positive duration response (Objective B). Establishing a positive duration response implies confirmation that cooling is effective in improving outcome or recovery versus normothermia, when a normothermia control arm is not clinically acceptable.

A maximal sample size of 1800 subjects enrolled over 4 years (estimated accrual rate of 37.5 subjects/month) is anticipated.

Investigational Device Exemption

ELIGIBILITY:
Inclusion Criteria:

* Coma after resuscitation from out of hospital cardiac arrest
* Cooled to <34 deg C with 240 minutes of cardiac arrest
* Definitive temperature control applied
* Age ≥ 18 years
* Informed consent from legal authorized representative (LAR) including intent to maintain life support for 96 hours
* Enrollment within 6 hours of initiation of cooling

Exclusion Criteria:

* Hemodynamic instability
* Pre-existing neurological disability or condition that confounds outcome determination
* Pre-existing terminal illness, unlikely to survive to outcome determination
* Planned early withdrawal of life support
* Presumed sepsis as etiology of arrest
* Prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1158 (Actual)
Dates: Start 2020-05-18 (Actual); Primary Completion 2025-09-05 (Estimated); Study Completion 2025-09-05 (Estimated)

PRIMARY OUTCOMES:
Weighted Modified Rankin Scale (mRS) | 90 days after return of spontaneous circulation
  The mRS is a 7 level ordinal scale of disability that ranges from 0 (no symptoms at all) to 6 (death). ICECAP uses weighting of mRS states to capture changes in functional status.

SECONDARY OUTCOMES:
All Cause Mortality | 90 days after return of spontaneous circulation
  All patients who are dead at follow up.
NIH Toolbox Crystallized Cognition Composite Score | 90 days after return of spontaneous circulation
  Composite T-scores from a subset of study neuropsychological tests evaluating.
NIH Toolbox Fluid Cognition Composite Score | 90 days after return of spontaneous circulation
  Composite T-scores from a subset of study neuropsychological tests evaluating cognitive functioning in awake survivors collected on the NIH Toolbox platform. The fluid cognition composite score is more reflective of capacity for new learning and information. processing in novel situations
Pneumonia | 90 days after return of spontaneous circulation
  Determined by simplified Centers for Disease Control and Prevention (CDC) National Healthcare Safety Network (NHSN) definitions of Ventilator-Associated Event (VAE) or Pneumonia.
Other infection | 90 days after return of spontaneous circulation
  Determined by simplified CDC NHSN (Center for Disease Control National Healthcare Safety Network) definitions of Urinary Tract Infection or Blood Stream Infection.
Malignant cardiac arrhythmia | 90 days after return of spontaneous circulation
  Defined as any arrhythmia that requires termination with chest compressions, pacing, defibrillation, or electrical cardioversion. Arrhythmias (including atrial fibrillation) managed only with medication are excluded.
Seizures | 90 days after return of spontaneous circulation
  Defined as unambiguous convulsive or electroencephalographic seizure activity triggering urgent initial or additional anticonvulsant therapy. This definition does not include those given further anticonvulsants as secondary prophylaxis or as treatment for vague or uncertain exam findings or nondiagnostic electroencephalography. It does not include myoclonus.
Neurological worsening | 90 days after return of spontaneous circulation
  Determined by a decrease in Full Outline of Unresponsiveness (FOUR) score of ≥4 points that persists on two consecutive days or is associated with a neurological death. It excludes transient fluctuations in neurological examination or changes attributed to pharmacological sedation or paralysis.
Electrolyte abnormalities | 90 days after return of spontaneous circulation
  Defined as a measured serum Na, K, Mg, or Ca that is either higher or lower than study defined boundaries on at least two sequential measurements and resulting in a change in IV therapy. It excludes deliberate hypernatremia or hypermagnesemia induced to treat intracranial hypertension or shivering.
Coagulopathies | 90 days after return of spontaneous circulation
  Defined as requiring all 3 of the following parameters: (1) some form of major bleeding associated with (2) laboratory confirmation of an abnormal clotting axis and (3) treatment with blood product transfusion or reversal agent. Laboratory testing may include International Normalized Ratio (INR), partial thromboplastin time (PTT), clotting time, or thromboelastography.

CONTACTS AND LOCATIONS:
Overall Officials: William Meurer, Principal Investigator — University of Michigan; Robert Silbergleit, Principal Investigator — University of Michigan; Romer Geocadin, Principal Investigator — Johns Hopkins University
Locations (76):
- United States (76):
  - University of Alabama Hospital, Birmingham, Alabama
  - Banner University Medical Center, Tucson, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Ronald Regan UCLA Medical Center, Los Angeles, California
  - UC Davis Medical Center, Sacramento, California
  - UC San Diego Medical Center - Hillcrest, San Diego, California
  - Zuckerberg San Francisco General Hospital, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - Harbor-UCLA Medical Center, Torrance, California
  - University of Colorado Hospital, Aurora, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - Yale New Haven Hospital, New Haven, Connecticut
  - George Washington University Hospital, Washington D.C., District of Columbia
  - UF Health Shands Hospital, Gainesville, Florida
  - Grady Memorial Hospital, Atlanta, Georgia
  - The Queen's Medical Center, Honolulu, Hawaii
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois-Chicago Hosptial, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - IU Health Methodist Hospital, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kentucky Hospital, Lexington, Kentucky
  - Maine Medical Center, Portland, Maine
  - University of Maryland Medical Center, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan Hospital, Ann Arbor, Michigan
  - Henry Ford Macomb Hospital, Clinton Township, Michigan
  - Detroit Receiving Hospital, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - DMC Sinai Grace Hospital, Detroit, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - M Health Fairview Southdale Hospital, Edina, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Cooper University Hospital, Camden, New Jersey
  - University of New Mexico, Albuquerque, New Mexico
  - South Shore University Hospital, Bay Shore, New York
  - NYU Langone Health - Tisch Hospital, New York, New York
  - The Mount Sinai Hospital, New York, New York
  - NYP Columbia University Medical Center, New York, New York
  - Strong Memorial Hospital, Rochester, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center, The Bronx, New York
  - Duke University Hospital, Durham, North Carolina
  - ECU Health Medical Center, Greenville, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - OSU East Hospital, Columbus, Ohio
  - OSU Wexner Medical Center, Columbus, Ohio
  - Mercy St. Vincent Medical Center, Toledo, Ohio
  - Adventist Health, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - UPMC Harrisburg, Harrisburg, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Guthrie Robert Packer Hospital, Sayre, Pennsylvania
  - Parkland Hospital, Dallas, Texas
  - Memorial Hermann Hospital, Houston, Texas
  - University of Utah Hospital, Salt Lake City, Utah
  - University of Virginia Medical Center, Charlottesville, Virginia
  - VCU Medical Center, Richmond, Virginia
  - Providence Regional Medical Center Everett, Everett, Washington
  - Harborview Medical Center, Seattle, Washington
  - Froedtert Hospital, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
The data will be stored in the NHLBI data repository after trial completion.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 1 year after publication on main outcome results paper
Access Criteria: Data use agreement with the appropriate NHLBI repository

REFERENCES:
- [Background] Meurer WJ, Schmitzberger FF, Yeatts S, Ramakrishnan V, Abella B, Aufderheide T, Barsan W, Benoit J, Berry S, Black J, Bozeman N, Broglio K, Brown J, Brown K, Carlozzi N, Caveney A, Cho SM, Chung-Esaki H, Clevenger R, Conwit R, Cooper R, Crudo V, Daya M, Harney D, Hsu C, Johnson NJ, Khan I, Khosla S, Kline P, Kratz A, Kudenchuk P, Lewis RJ, Madiyal C, Meyer S, Mosier J, Mouammar M, Neth M, O'Neil B, Paxton J, Perez S, Perman S, Sozener C, Speers M, Spiteri A, Stevenson V, Sunthankar K, Tonna J, Youngquist S, Geocadin R, Silbergleit R; ICECAP trial investigators. Influence of Cooling duration on Efficacy in Cardiac Arrest Patients (ICECAP): study protocol for a multicenter, randomized, adaptive allocation clinical trial to identify the optimal duration of induced hypothermia for neuroprotection in comatose, adult survivors of after out-of-hospital cardiac arrest. Trials. 2024 Jul 23;25(1):502. doi: 10.1186/s13063-024-08280-w. PMID 39044295
- [Derived] Meurer W, Schmitzberger F, Yeatts S, Ramakrishnan V, Abella B, Aufderheide T, Barsan W, Benoit J, Berry S, Black J, Bozeman N, Broglio K, Brown J, Brown K, Carlozzi N, Caveney A, Cho SM, Chung-Esaki H, Clevenger R, Conwit R, Cooper R, Crudo V, Daya M, Harney D, Hsu C, Johnson NJ, Khan I, Khosla S, Kline P, Kratz A, Kudenchuk P, Lewis RJ, Madiyal C, Meyer S, Mosier J, Mouammar M, Neth M, O'Neil B, Paxton J, Perez S, Perman S, Sozener C, Speers M, Spiteri A, Stevenson V, Sunthankar K, Tonna J, Youngquist S, Geocadin R, Silbergleit R. Influence of Cooling duration on Efficacy in Cardiac Arrest Patients (ICECAP): study protocol for a multicenter, randomized, adaptive allocation clinical trial to identify the optimal duration of induced hypothermia for neuroprotection in comatose, adult survivors of after out-of-hospital cardiac arrest. Res Sq [Preprint]. 2024 Jun 21:rs.3.rs-4033108. doi: 10.21203/rs.3.rs-4033108/v1. PMID 38947064
- [Derived] Chen CT, Lin JW, Wu CH, Kuo RN, Shih CH, Hou PC, Yen DH, How CK. A Simple Risk Score for Predicting Neurologic Outcome in Out-of-Hospital Cardiac Arrest Patients After Targeted Temperature Management. Crit Care Med. 2022 Mar 1;50(3):428-439. doi: 10.1097/CCM.0000000000005266. PMID 34495880

DOCUMENTS (2):
  • Study Protocol (2020-05-04): https://cdn.clinicaltrials.gov/large-docs/51/NCT04217551/Prot_000.pdf
  • Informed Consent Form (2020-05-04): https://cdn.clinicaltrials.gov/large-docs/51/NCT04217551/ICF_001.pdf